CLINICAL TRIAL: NCT03371004
Title: A Phase I Trial to Evaluate Safety and Tolerance of Intravenous 4-Demethyl-4-cholesteryloxycarbonylpenclomedine (DM-CHOC-PEN) in Adult Subjects With Cancer Involving the CNS
Brief Title: DM-CHOC-PEN Plus Radiation for Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DEKK-TEC, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DTI-025
Record Dates: First submitted 2017-11-19; First posted 2017-12-13 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Advanced Cancer
Keywords: DM-CHOC-PEN; Radiation; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DM-CHOC-PEN + Radiation (Experimental): 4-Demethyl-4-cholesteryloxycarbonylpenclomedine (DM-CHOC-PEN) - 39-89.7 MG/M2 iv once and then 3-weeks later radiation - 15-30 Gy will be administered
  Interventions: Drug: 4-Demethyl-4-cholesteryloxycarbonylpenclomedine

INTERVENTIONS:
Drug: 4-Demethyl-4-cholesteryloxycarbonylpenclomedine — IV administration as described
  Other Names: DM-CHOC-PEN

SUMMARY:
4-Demethyl-4-cholesteryloxycarbonylpenclomedine (DM-CHOC-PEN) is a polychlorinated pyridyl cholesterol carbonate that is lipophilic, electrically neural, crosses the blood brain barrier (BBB), ability to localize in intracranial tumor tissue, lacks neurotoxicity and not transported out of the brain via Pgp (p-glycoprotein) (1). DM-CHOC-PEN has completed Phase I/II trials in humans with primary and secondary tumors involving the brain with success. Complete remissions in both primary astrocytoma and metastatic lung and leukemia malignancies.

This trial is open for adult subjects with advanced cancer - brain involvement is required.

DETAILED DESCRIPTION:
The primary goal of this Phase I oncology clinical trial will be to evaluate the safety and use of 4-demethyl-4-cholesteryloxycarbonylpenclomedine (DM-CHOC-PEN) plus radiation, as anticancer therapy for adults with advanced cancer involving the central nervous system (CNS) involvement.

DM-CHOC-PEN is a polychlorinated pyridine cholesteryloxycarbonate that crosses the blood brain barrier (BBB), accumulates in CNS tumor tissue in humans and has produced objective responses, with acceptable/reversible hepatic toxicities (in patients with prior liver disease) and no evidence of hematological, renal, neuro-toxicities with improved quality of life and overall survival in adult Phase I/II clinical trials - IND - 68,876.

The drug recently received Orphan Drug designation for NSCLC involving the brain.

The FDA supports the proposed Phase I clinical trial designed to identify safety, toxicities and an acceptable MTD of the drug in combination with radiation in adult cancers subjects with CNS involvement.

Almost 700,000 people in the US are living with tumors involving the CNS or spinal nervous system (SNS) tumors. Trends in CNS tumors have sharply increased since 1989 for individuals with a history of cancer, who appeared to have 'beaten the odds', only to have a reoccurrence from cancer involving the CNS after years of remission; the most common types of cancer in AYA individuals are - from lung, breast, melanoma, and sarcoma malignancies. This group of individuals deserves special attention.

A critical component in designing an agent that will cross the protective blood brain barrier (BBB) is that the agent must be readily transported intracerebrally, does not produce local irritation/neurotoxicity and is not recycled back into the general circulation. After IV administration DM-CHOC-PEN readily penetrates the BBB, is not a substrate for the transporter protein P-glycoprotein (P-gp) and has shown anticancer activity in CNS tumors. The effective transport of DM-CHOC-PEN into CNS tumors in adults without neurotoxic behavioral alterations and associated events supports the drug's use in combination with radiation in the treatment of CNS tumors. The observed responses noted in adults with metastatic cancers involving the CNS and cerebellum treated with DM-CHOC-PEN is encouraging. Thus, the drug's unique properties and lack of toxicities noted in the adult studies merits the Phase I trial proposed here in combination with radiation.

The specific objectives of this Phase I study will be to:

1. Conduct a Phase I clinical trial with DM-CHOC-PEN plus radiation in adults with advanced cancers involving the central nervous system to document toxicities, define an acceptable maximum tolerated dose (MTD), and identify anticancer activity for the binary treatment DM-CHOC-PEN plus radiation. All data will be communicated through an e-RAP program. This will be accomplished through IND - 68.876.
2. Studying the pharmacokinetic/dynamic profiles of DM-CHOC-PEN and metabolites in adults after being treated with DM-CHOC-PEN and radiation.
3. Analyze data and prepare a Phase II clinical trial or a Designation Orphan Drug application for FDA review.

ELIGIBILITY:
Inclusion Criteria:: Inclusion Criteria will be as follows -

* Subjects must have histological proof of a CNS malignancy (primary or metastatic), which has been treated with standard treatments, that may include radiation, and must have measurable lesions.
* Subjects must have life expectancy of at least 12 weeks and a Karnofsky performance score: > 60 % (or a Zubrod performance status of < 2).
* The age limit - a limit of 39 years of age. Gender is not a criterion.
* All subjects must be off previous chemo- and/or radiotherapy for at least three (3) weeks prior to entrance into the study and have recovered from any toxic effects induced by such treatment(s); no nitrosourea type drug or ipilumimab treatments are permitted within the last six (6) weeks prior to enrollment. No major surgery within 14 days of enrollment. Subjects may continue to receive anti- estrogen/steroid therapy that has been initiated at least eight weeks prior to enrollment in the study.
* Subjects should have adequate bone marrow function defined as a peripheral WBC >3,000/mm3 with an ANC >1500/mm3 and a platelet count >100,000/mm3.
* Subjects should have hepatic function (alkaline phosphatase, AST and ALT) < ULN and renal functions with serum creatinine - <1.5 x UNL. If a patient has liver metastasis and/or a history of liver disease - they will receive a lower dose of the drug per treatment protocol.
* Subjects should not be allergic to eggs or soy beans.
* Subjects must be medically, psychologically and neurologically stable and have triplicate baseline ECG's with a mean QTc interval <500 ms and >300 ms and neither a history of congenital prolonged or short QT syndrome. Subjects with a history of cardiac disease must be stable.
* Subjects and/or legal guardian must understand the nature of the study and be willing to sign an informed consent that complies with the investigator/DEKK-TEC policies and approved by the Human Investigation Review Committee.

Exclusion Criteria:Criteria: Inclusion Criteria: Inclusion Criteria will be as follows -

* Subjects must have histological proof of a CNS malignancy (primary or metastatic), which has been treated with standard treatments, that may include radiation, and must have measurable lesions.
* Subjects must have life expectancy of at least 12 weeks and a Karnofsky performance score: > 60 % (or a Zubrod performance status of < 2).
* The age limit - a limit of 39 years of age. Gender is not a criterion.
* All subjects must be off previous chemo- and/or radiotherapy for at least three (3) weeks prior to entrance into the study and have recovered from any toxic effects induced by such treatment(s); no nitrosourea type drug or ipilumimab treatments are permitted within the last six (6) weeks prior to enrollment. No major surgery within 14 days of enrollment. Subjects may continue to receive anti- estrogen/steroid therapy that has been initiated at least eight weeks prior to enrollment in the study.
* Subjects should have adequate bone marrow function defined as a peripheral WBC >3,000/mm3 with an ANC >1500/mm3 and a platelet count >100,000/mm3.
* Subjects should have hepatic function (alkaline phosphatase, AST and ALT) < ULN and renal functions with serum creatinine - <1.5 x UNL. If a patient has liver metastasis and/or a history of liver disease - they will receive a lower dose of the drug per treatment protocol.
* Subjects should not be allergic to eggs or soy beans.
* Subjects must be medically, psychologically and neurologically stable and have triplicate baseline ECG's with a mean QTc interval <500 ms and >300 ms and neither a history of congenital prolonged or short QT syndrome. Subjects with a history of cardiac disease must be stable.
* Subjects and/or legal guardian must understand the nature of the study and be willing to sign an informed consent that complies with the investigator/DEKK-TEC policies and approved by the Human Investigation Review Committee.

Exclusion Criteria: Exclusion criteria will be as follows:

* Subjects with concurrent severe and/or uncontrolled medical co-morbidities - including active infections, unstable uncontrolled diabetes, cardiovascular and pulmonary, renal, psychiatric or social conditions that could compromise the safety or compliance of treatment are not eligible.
* Concomitant chemotherapy or radiotherapy is not permitted.
* Pregnant or lactating females are excluded. Women of childbearing age, and their sexual partners, must use an effective contraception program. Males who are having sexual relations with women capable of child bearing must use the barrier birth control while on the study and for 3-months after the last dose of the study drug.
* Subjects taking CYP3A4 inducers or inhibitors are not eligible since it is not known whether the study drug is metabolized through this pathway. The following CYP3A4 inhibitors/inducers are not permitted during the trial - phenobarbital, fluconazole, erythromycin, verapamil; the latter 3-drugs are moderate CYP3A4 inhibitors.
* Subjects taking the following medications may experience QT/QTc interval prolongation and are not eligible for the trial - most anti-arrhythmia drugs (incl. amiodarone), erythromycin, quinolone antibiotics, ketoconazole, Zithromax, and phenothiazine and will be denied enrollment in the study. The possible interactions of these drugs and DM-CHOC-PEN have not been established. Subjects receiving these drugs will only be eligible if they discontinue the drugs and have an acceptable ECG.
* Coagulopathies - patients requiring full dose anticoagulation with warfarin are excluded. However, patients stable and on other anticoagulants can be incl

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-02-05 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 year
  Laboratory and imaging studies to verify responses

SECONDARY OUTCOMES:
Imaging studies | 6-weeks after treatments
  MRI Exams of the Brain after Treatments

CONTACTS AND LOCATIONS:
Overall Officials: Steven DiBiase, MD, Principal Investigator — Tulane University Medical Center; Lee Roy Morgan, MD, PhD, Principal Investigator — DEKK-TEC, Inc.
Locations (3):
- United States (3):
  - Tulane University Medical Center, New Orleans, Louisiana
  - Tulane University Medical School, New Orleans, Louisiana
  - Detroit Clinical Research Centers, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: Yes
Other trial centers are being evaluated
Supporting Information: Study Protocol, ICF
Time Frame: Upon release of the Clinical Trials.gov approval
URL: http://dekk-tec.com